CLINICAL TRIAL: NCT01867424
Title: Pilot Study of Eovist (Gadoxetate) Enhanced MRI for the Detection of Prostate Cancer
Brief Title: Gadoxetate Enhanced Imaging Study to Detect Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ismail B. Turkbey, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 130145; 13-C-0145
Record Dates: First submitted 2013-05-31; First posted 2013-06-04 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: Testosterone Membrane Transporter; OATP1B3; Castration Resistant Prostate Cancer; Prostatectomy; Gadolinium-Based Contrast Agent
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with Advanced Disease (Active Comparator): Advanced disease: who have failed hormone therapy and who have sufficient tissue from a soft tissue or metastatic bone lesion (measuring 1.5cm in diameter at computed tomography (CT) or magnetic resonance imaging (MRI) scan) available for organic anion-transporting polypeptide 1B3 (OATP1B3) immunohistochemistry (IHC) or must have a soft tissue or metastatic bone lesion that can be biopsied and be willing to undergo percutaneous biopsy to obtain tissue for OATP1B3 expression.
  Interventions: Drug: Eovist
- Participants with Localized Disease (Active Comparator): Localized disease: must have image guided biopsy confirmed prostate cancer and sufficient tissue available for OATP1B3 IHC.
  Interventions: Drug: Eovist

INTERVENTIONS:
Drug: Eovist — 0.1 ml/kg Eovist will be administered intravenous (IV) to each patient

SUMMARY:
Background:

- Prostate cancer is the most common cancer type among men. Some prostate cancers respond to hormonal therapy. However, some cell characteristics of other prostate cancers cause it not to respond as well to these therapies. Researchers want to see if gadoxetate, a contrast agent used to help identify damaged liver tissue, can help tell these types of prostate cancer apart. It may be able to identify if a man has a type of prostate cancer for which hormone therapy may not work as well.

Objectives:

- To see if gadoxetate can help identify different types of prostate cancers during imaging studies.

Eligibility:

- Men at least 18 years of age who have prostate cancer. Participants will be having surgery to either remove the prostate or take tumor tissue samples.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected.
* Participants will have a magnetic resonance imaging (MRI) scan of the lower torso. They will receive gadoxetate during the MRI scan.
* Participants who have surgery will have a sample of their tumor cells collected. Those who have a biopsy will provide cells from this biopsy for study.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
BACKGROUND:

* Prostate cancer is the most common non-cutaneous malignancy among men in the western world. Prognostic biomarkers would be useful in stratifying patients to different treatments.
* The expression of a testosterone membrane transporter, organic anion-transporting polypeptide 1B3 (OATP1B3), is associated with shorter time to progression after hormonal ablation therapy and shorter overall survival in prostate cancer patients. 52% of localized prostate cancer lesions express OATP1B3, while 92% of prostate cancer metastases requiring hormonal ablation treatment, express OATP1B3 in soft tissue lesions. Expression of OATP1B3 also correlates with Gleason grade.
* Current imaging methods cannot predict treatment failure or resistance.
* Gadoxetate disodium (Gd-EOB-DTPA) (Eovist , Bayer HealthCare Pharmaceuticals Inc. Pittsburgh, PA) is an MR imaging agent which is FDA-approved gadolinium chelate for detecting hepatocellular carcinoma (HCC), as normal hepatocytes express OATP1B3 while most hepatocellular carcinomas (HCC) do not. However, those HCCs that do take up Eovist have been shown to express OATP1B3.
* Eovist may be useful to evaluate OATP1B3 status in patients with prostate cancer and may therefore serve as a prognostic and treatment biomarker.

PRIMARY OBJECTIVE:

-Evaluate the uptake and retention of Eovist in prostate cancers.

ELIGIBILTY:

* Male subjects greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2
* Subjects with clinically localized prostate cancer must have image guided biopsy confirmed prostate cancer and sufficient tissue available for OATP1B3 immunohistochemistry (IHC).
* Subjects with advanced disease who have failed hormone therapy and who have sufficient tissue from a soft tissue or metastatic bone lesion (measuring greater than or equal to1.5cm in diameter at computed tomography (CT) or magnetic resonance imaging (MRI) scan) available for OATP1B3 IHC.

or

-Subjects, for whom tissue is not available, must have a soft tissue or metastatic bone lesion that can be biopsied and be willing to undergo percutaneous biopsy to obtain tissue for OATP1B3 expression.

DESIGN:

* This pilot study will accrue 25 subjects divided into two arms: 10 evaluable subjects with localized prostate cancer and 15 evaluable subjects with advanced disease
* Each subject will receive a single intravenous (IV) dose of Eovist by bolus injection
* All subjects will undergo magnetic resonance imaging (MRI) prior to and immediately after, 10, 20 and 60 minutes post-Eovist injection

ELIGIBILITY:
* INCLUSION CRITERIA:

2.1.1.1 Subject is greater than or equal to 18 years old.

2.1.1.2 Subjects with clinically localized prostate cancer (outside pathology is acceptable) must have image guided biopsy confirmed prostate cancer and sufficient tissue available (obtained before or after 20 weeks of Eovist injection) for organic anion-transporting polypeptide 1B3 (OATP1B3) expression.

2.1.1.3 Subjects with advanced disease who have failed hormone therapy and who have sufficient tissue (obtained before or after 20 weeks of Eovist injection) from a soft tissue lesion (measuring greater than or equal to 1.5cm in diameter at computed tomography (CT) or magnetic resonance imaging (MRI) scan) available for OATP1B3 expression.

or

2.1.1.4 Subjects, for whom tissue is not available, must have a soft tissue or metastatic bone lesion that can be biopsied and be willing to undergo percutaneous biopsy to obtain tissue for OATP1B3 expression.

2.1.1.5 Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

2.1.1.6 Serum creatinine within 3 weeks prior to Eovist MRI less than or equal to 1.8mg/dl and estimated glomerular filtration rate (eGFR) must be greater than 30 ml/min/1.73m(2).

2.1.1.7 Patients must have normal liver function as defined below:

* total bilirubin less than 2 times normal institutional limits or greater than 3.0 mg/dl in patients with Gilberts syndrome
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 times institutional upper limit of normal

2.1.1.8 Ability of subject to sign a written informed consent document

EXCLUSION CRITERIA:

2.1.2.1 Subjects with known hypersensitivity and allergy to gadolinium contrast agents

2.1.2.2 Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results

2.1.2.3 Subjects with severe claustrophobia unresponsive to oral anxiolytics

2.1.2.4 Subjects with contraindications to magnetic resonance imaging (MRI)

2.1.2.5 Subjects weighing greater than 136 kg (weight limit for scanner table)

2.1.2.6 Subjects with pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI

2.1.2.7 Subjects with other medical conditions deemed by the principle investigator (or associates) to make the subject ineligible for protocol procedures

2.1.2.8 Subjects who will have a delay in clinically indicated radiation therapy due to the interval between Eovist MRI imaging and biopsy

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 2.1.1.1 Subject is greater than or equal to 18 years old.
  2.1.1.2 Subjects with clinically localized prostate cancer (outside pathology is acceptable) must have image guided biopsy confirmed prostate cancer and sufficient tissue available (obtained before or after 20 weeks of Eovist injection) for organic anion-transporting polypeptide 1B3 (OATP1B3) expression.
  2.1.1.3 Subjects with advanced disease who have failed hormone therapy and who have sufficient tissue (obtained before or after 20 weeks of Eovist injection) from a soft tissue lesion (measuring greater than or equal to 1.5cm in diameter at computed tomography (CT) or magnetic resonance imaging (MRI) scan) available for OATP1B3 expression.
  or
  2.1.1.4 Subjects, for whom tissue is not available, must have a soft tissue or metastatic bone lesion that can be biopsied and be willing to undergo percutaneous biopsy to obtain tissue for OATP1B3 expression.
Enrollment: 24 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismail B Turkbey, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narita M, Hatano E, Arizono S, Miyagawa-Hayashino A, Isoda H, Kitamura K, Taura K, Yasuchika K, Nitta T, Ikai I, Uemoto S. Expression of OATP1B3 determines uptake of Gd-EOB-DTPA in hepatocellular carcinoma. J Gastroenterol. 2009;44(7):793-8. doi: 10.1007/s00535-009-0056-4. Epub 2009 Apr 29. PMID 19404564
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Hamada A, Sissung T, Price DK, Danesi R, Chau CH, Sharifi N, Venzon D, Maeda K, Nagao K, Sparreboom A, Mitsuya H, Dahut WL, Figg WD. Effect of SLCO1B3 haplotype on testosterone transport and clinical outcome in caucasian patients with androgen-independent prostatic cancer. Clin Cancer Res. 2008 Jun 1;14(11):3312-8. doi: 10.1158/1078-0432.CCR-07-4118. PMID 18519758
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0145.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Advanced Disease | Participants With Localized Disease
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1
Not completed — Patient noncompliance | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Advanced Disease | Participants With Localized Disease | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.67 (10.59) | 65.17 (7.30) | 65.42 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Uptake and Retention of Eovist in Prostate Cancers
Description: Uptake and retention of Eovist in prostate cancers is measured by the change of magnetic resonance imaging (MRI) parameter values between pre and post injection.
Time Frame: Baseline and 20 minutes, 40 minutes, and 60 minutes after Eovist injection
Population: Three patients did not complete the study and are excluded, and two patients were not evaluable due to non-evaluable images.
Measure: Mean (Standard Deviation); unit: contrast enhancement ratio (CER)
Arm/Group | Participants With Advanced Disease | Participants With Localized Disease
Number analyzed (Participants) | 9 | 10
contrast enhancement ratio (CER)
  Baseline | 2.01 (1.16) | 1.857 (0.41)
  20 minutes after Eovist | 2.52 (1.26) | 2.212 (0.36)
  40 minutes after Eovist | 2.52 (1.39) | 2.05 (0.34)
  60 minutes after Eovist | 2.56 (1.45) | 2.06 (0.34)
Statistical Analysis 1: Comparison: Participants With Advanced Disease vs Participants With Localized Disease; Null Hypothesis: There is no significant difference in contrast enhancement ratio (CER) in prostate cancers upon injection of Eovist. Subgroup analysis of CER in (i) Advanced Disease and (ii) Localized Disease; Test type: Other; p = 0.0008, Wilcoxon Test — Median of difference in CER: All cases; Median of Differences = 0.43 — The relative difference between groups is based on the change from baseline values to the values collected at each of the three time points
Statistical Analysis 2: Comparison: Participants With Advanced Disease; Test type: Other; p = 0.0039, Wilcoxon Test — Median of difference in CER: Advanced Disease Cases; Median of Differences = 0.42
Statistical Analysis 3: Comparison: Participants With Localized Disease; Test type: Other; p = 0.084, Wilcoxon Test — Median of difference in CER: Local Disease Cases; Median of Differences = 0.475
Statistical Analysis 4: Comparison: Participants With Localized Disease; Analysis of CER from baseline to 40 minutes after Eovist injection; Test type: Other; p = 0.25, Wilcoxon Test; Median Difference CER = 0.17
Statistical Analysis 5: Comparison: Participants With Localized Disease; Analysis of CER from baseline to 60 minutes after Eovist injection; Test type: Other; p = 0.1602, Wilcoxon Test; Median Difference CER = 0.27
Statistical Analysis 6: Comparison: Participants With Advanced Disease; Analysis of CER from baseline to 40 minutes after Eovist injection; Test type: Other; p = 0.0078, Wilcoxon Test; Median Difference CER = 0.29
Statistical Analysis 7: Comparison: Participants With Advanced Disease; Analysis of CER from baseline to 60 minutes after Eovist injection; Test type: Other; p = 0.0039, Wilcoxon Test; Median Difference CER = 0.34
Statistical Analysis 8: Comparison: Participants With Advanced Disease vs Participants With Localized Disease; Analysis of CER from baseline to 40 minutes after Eovist injection; Total cases; Test type: Other; p = 0.0046, Wilcoxon Test; Median Difference CER = 0.27
Statistical Analysis 9: Comparison: Participants With Advanced Disease vs Participants With Localized Disease; Analysis of CER from baseline to 60 minutes after Eovist injection; Total cases; Test type: Other; p = 0.0017, Wilcoxon Test; Median Difference CER = 0.33

2. Secondary Outcome: Number of Participants Who Were Evaluated for Magnetic Resonance (MR) Contrast Enhancement Parameters Following Eovist Injection With Respect to Gleason Score
Description: Scans with or without endorectal coil were obtained through the prostate gland, bone metastasis or soft tissue metastasis (usually a lymph node) selected as the target lesion as described in primary outcome measure. Then 0.1 ml/kg Eovist was administered intravenously. Scans were correlated with baseline Gleason score obtained from the prostate biopsy. Gleason score <7 = low grade cancer; Gleason score ≥7 = high grade cancer.
Time Frame: At baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Advanced Disease | Participants With Localized Disease
Number analyzed (Participants) | 9 | 10
Participants
  Gleason score <7 | 0 | 1
  Gleason score ≥7 | 9 | 9

3. Secondary Outcome: Baseline Serum Prostate-Specific Antigen (PSA) Levels of Patients Who Were Evaluated for Magnetic Resonance (MR) Contrast Enhancement Parameters Following Eovist Injection
Description: Scans with or without endorectal coil were obtained through the prostate gland, bone metastasis or soft tissue metastasis (usually a lymph node) selected as the target lesion as described in primary outcome measure. Then 0.1 ml/kg Eovist was administered intravenously. Scans were correlated to baseline PSA levels.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Advanced Disease | Participants With Localized Disease
Number analyzed (Participants) | 9 | 10
ng/mL | 163.17 (208.50) | 11.46 (13.15)
Statistical Analysis 1: Comparison: Participants With Advanced Disease vs Participants With Localized Disease; Null Hypothesis: There is no significant difference in contrast enhancement ratio (CER) with Eovist injection based on baseline Prostate-specific antigen (PSA) levels at 20-minute timepoint; Test type: Other; p = 0.5761, Nonparametric Spearman correlation; The calculation of Spearman correlation is between baseline PSA and CER at 20 minutes post Eovist injection; Spearman r = -0.1370, 95% CI 2-sided [-0.5665 to 0.3511]
Statistical Analysis 2: Comparison: Participants With Advanced Disease vs Participants With Localized Disease; Analyses include calculation of Spearman correlation between baseline Prostate-specific antigen (PSA) and CER at 40 minutes post Eovist injection; Test type: Other; p = 0.3033, nonparametric Spearman correlation; Spearman r = -0.2570, 95% CI 2-sided [-0.6549 to 0.2526]
Statistical Analysis 3: Comparison: Participants With Advanced Disease vs Participants With Localized Disease; Analyses include calculation of Spearman correlation between baseline Prostate-specific antigen (PSA) and CER at 60 minutes post Eovist injection; Test type: Other; p = 0.2351, nonparametric Spearman correlation; Spearman r = -0.2861, 95% CI 2-sided [-0.6634 to 0.2071]
Statistical Analysis 4: Comparison: Participants With Localized Disease; Analyses include analysis of CER at 20 minutes after Eovist injection based on baseline Prostate-specific antigen (PSA) stratifying by PSA < or >/= 20ng/ml; Test type: Other; p = 0.111, Mann Whitney; Median Difference (actual) = -0.47
Statistical Analysis 5: Comparison: Participants With Advanced Disease; [analysis description as in outcome 3, analysis 4]; Test type: Other; p = 0.7738, Mann Whitney; Median Difference (actual) = -0.7750

4. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From date treatment consent signed to date off study, approximately 3 years and 33 days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Advanced Disease | Participants With Localized Disease
Number analyzed (Participants) | 12 | 12
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From date treatment consent signed to date off study, approximately 3 years and 33 days
Arm/Group | Participants With Advanced Disease | Participants With Localized Disease
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Advanced Disease (N=12) | Participants With Localized Disease (N=12)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-05-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT01867424/Prot_SAP_ICF_000.pdf